CLINICAL TRIAL: NCT04460417
Title: Health Behavior and Feedback Among Chicago Area Communities
Brief Title: Chicago Community Health Study
Acronym: CCHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1573
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced care (Experimental): Participants will take part in an approximate one-hour health and smoking feedback session at the University of Chicago in Dr. King's Clinical Addictions Research Laboratory (CARL). The session will follow the Courage to Quit™ (CTQ) Roadmap program (developed by Dr. King with the Respiratory Health Association). This roadmap shorter version of the larger CTQ program has been specifically designed as an inpatient bedside or outpatient brief intervention guide to assess smoking cessation motivation, consequences of smoking, facts and myths about smoking, barriers to making a change, approved medications, de-bunking myths about medications or treatments without scientific evidence (e-cigarette, laser treatments, herbals, etc.), and gaining social support.
  Interventions: Behavioral: Enhanced Care
- Treatment as Usual (Active Comparator): Participants will receive the National Cancer Institute (NCI) pamphlet "Clearing the Air" and access to related online resources, which includes brief advice to quit smoking and medication information.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Enhanced Care — The session began with the therapist reviewing the participants' personal feedback sheet within the context of clear messaging that there is no safe level of smoking and of how smoking affects the participant individually and the Black community collectively. The participant was encouraged to quit smoking, else to reduce smoking if abstinence was not desired, and to use NRT within the next week to help foster behavior change and alleviate withdrawal symptoms. This portion of the counseling was presented within a culturally-targeted framework such that myths regarding NRT common among persons with low health literacy were discussed and debunked and historical mistrust of the medical community and concerns about exploitation were also addressed. Each participant in EC was offered a starter kit of NRT with a one week supply of patches or lozenges.
  Other Names: EC
  Arms: Enhanced care
Behavioral: TAU — Participants met with a research assistant for 3-5 minutes and received the National Cancer Institute (NCI) pamphlet "Clearing the Air" and access to related online resources, which includes brief advice to quit smoking and medication information. They did not receive counseling or specialized care and were advised to refer to the resources should they be interested in quitting smoking.
  Arms: Treatment as Usual

SUMMARY:
The study examined smokers from the initial COMPASS survey who live in one of three local Census tracks with large concentrations of minority populations and smoking rates, including Washington Park (98.8% African American, 60.5% smoker), Gage Park (76.7% Hispanic, 26.7% smoker), and Bridgeport (34.5% Asian, 27.0% Hispanic, 29.3% smoker), randomizing them to receipt of treatment as usual care advice (via a pamphlet form the National Cancer Institute) versus theoretically-driven and empirically-supported smoking cessation advice session delivered in-person at the UCM.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in either the Washington Park, Gage Park, or Bridgeport communities based on current physical address at the time of initial contact for study participation
* Identify as a current smoker (verified by self-report and exhaled carbon monoxide)
* Willing and able to sign an informed consent
* Stable residence and contact information throughout the follow-up period

Exclusion Criteria:

* Not a current smoker
* Does not live within the pre-determined neighborhood locations
* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Smoking reduction | Past-week CPD at 1- and 6-month follow-up
  Change in average cigarettes per day (CPD)
Quit attempts | Any reported (and serious) quit attempts since last session at 1- and 6-month follow-up
  Change in number of any and serious (12+hr) quit attempts
Motivation to change smoking | Increases in stage of change at 1- and 6-month follow-ups
  Increase in motivation to change smoking behavior via smoking contemplation ladder (Biener-Abrams Contemplation Ladder) scores. Scores are on a 10-point scale from 0-10, with higher scores indicating higher motivation to quit smoking.
Nicotine Replacement Therapy (NRT) use | Any reported NRT use since last session at 1- and 6- month follow-up
  Change in frequency of NRT use
Nicotine Replacement Therapy (NRT) knowledge | More accurate knowledge about NRT at 1- and 6-month follow-ups
  Increase in accurate knowledge about NRT assessed by two items rated from a 1 (strongly disagree) to 7 (strongly agree) scale measuring agreement to the NRT myths, "NRT causes cancer" and "NRT is only used by weak people".

CONTACTS AND LOCATIONS:
Overall Officials: Andrea King, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brett EI, Chavarria J, Liu M, Hedeker D, King AC. Effects of a brief motivational smoking intervention in non-treatment seeking disadvantaged Black smokers. J Consult Clin Psychol. 2021 Apr;89(4):241-250. doi: 10.1037/ccp0000629. Epub 2021 Mar 11. PMID 33705158